CLINICAL TRIAL: NCT00319345
Title: Sodium-Lactate Versus Mannitol in the Treatment of Intracranial Hypertensive Episodes in Severe Traumatic Brain Injured Patients
Brief Title: Sodium-Lactate and Traumatic Brain Injury
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institut d'Anesthesiologie des Alpes Maritimes (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); PT Kalbe Farma Tbk (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CHUN-LM-0001
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2006-04

CONDITIONS: Severe Trauma Brain Injury; Intracranial Hypertension
Keywords: Traumatic brain injury; Intracranial pressure; Osmotherapy; Glasgow outcome score; Mannitol; Sodium-Lactate
MeSH Terms: conditions — Intracranial Hypertension; Brain Injuries, Traumatic | interventions — Mannitol; Sodium Lactate

INTERVENTIONS:
Drug: Mannitol, Sodium-Lactate

SUMMARY:
The purpose of this study is to compare the effect of bolus of either sodium-lactate or mannitol on the evolution of intracranial pressure (ICP) during intracranial hypertensive episodes (IHE)

DETAILED DESCRIPTION:
Osmotherapy with mannitol remains the first treatment currently recommended to treat intracranial hypertension in severe head injury.However, this treatment in not always efficient and is associated with side-effects and a transitory action. Hypertonic sodium-lactate, by its osmotic and energetic properties could be superior to mannitol to decrease ICP. Study objectives : to compare the effect of mannitol and sodium-lactate on ICP at the fourth hour after the start of infusion during IHE in severe traumatic brain injury (TBI) (main endpoint) ; to compare the percentage of successfully treated episodes between both treatments and to compare the neurological status after one year of evolution (glasgow outcome score)(secondary endpoints)

Patients inclusion : adult severe TBI (glasgow coma score < 9) < 66 yrs Exclusion criteria : polytrauma, bilateral fixed dilated pupils, motor score < 4, neurosurgery, prolonged episode of hypoxia or arterial hypotension, 34 patients included from november 2003 to november 2004 and randomized into two groups : MAN group receiving mannitol 20% 100 ml in 15 min (17 patients, 36 episodes of IHE treated) and LAC group receiving semimolar sodium-lactate 100 ml in 15 min (17 patients, 37 episodes of IHE treated). For ethical reasons a rescue treatment in a crossover fashion was performed for each episode of IHE when the randomized treatment failed.

Follow-up : one year after the TBI. Study end : november 30, 2005

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years
* severe traumatic brain injury
* prehospital glasgow coma scale < 9
* rapid neurological worsening before admission

Exclusion Criteria:

* neurosurgical intervention
* polytrauma
* bilatéral fixed dilated pupils
* motorscore < 4
* prolonged episode of hypoxia or arterial hypotension
* abundant rinorrhea

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34
Dates: Start 2003-11; Study Completion 2005-11

PRIMARY OUTCOMES:
Efficiency to decrease ICP during IHE episodes

SECONDARY OUTCOMES:
Number of successful treatment, neurological status (Glasgow outcome score) after one year of evolution

CONTACTS AND LOCATIONS:
Overall Officials: Carole R ICHAI, MD-PhD, Study Director
Locations (1):
- CHU de Nice, Nice, Alpes Maritimes, France